CLINICAL TRIAL: NCT07360717
Title: To Compare the Efficacy & Safety of Ultra-Slow (24 hr) Low Dose (25 mg) Infusion of Alteplase Over Slow (24hr) Infusion of Streptokinase in Mechanical Prosthetic Valve Thrombosis : A Randomized Controlled Trial
Brief Title: To Compare the Efficacy & Safety of Ultra-Slow (24 hr) Low Dose (25 mg) Infusion of Alteplase Over Slow (24hr) Infusion of Streptokinase in Mechanical Prosthetic Valve Thrombosis
Acronym: PHVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: U. N. Mehta Institute of Cardiology and Research Center (Other)
Responsible Party: Principal Investigator, Dr. Sibasis Sahoo, Professor, Department of Cardiology, U. N. Mehta Institute of Cardiology and Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHVT
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Thrombolysed
Keywords: Pulmonary heart valve thrombosis
MeSH Terms: interventions — Tissue Plasminogen Activator; Streptokinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alteplase (Active Comparator): Low Dose (25 mg) Ultra-slow (24 hr) Infusion of Alteplase Without Bolus (max 72 hrs)
  Interventions: Drug: Alteplase; Drug: streptokinase
- Streptokinase (Active Comparator): Slow (24hr) Infusion of 25 lac units Streptokinase (2.5 lac 1st hr → 1 lac /hr for 23 hrs) (max 48 hrs)
  Interventions: Drug: Alteplase; Drug: streptokinase

INTERVENTIONS:
Drug: Alteplase — Low Dose (25 mg) Ultra-slow (24 hr) Infusion of Alteplase Without Bolus (max 72 hrs)
Drug: streptokinase — Slow (24hr) Infusion of 25 lac units Streptokinase (2.5 lac 1st hr → 1 lac /hr for 23 hrs) (max 48 hrs)

SUMMARY:
Annual incidence of PVT for mechanical valves is 0.3 - 1.3% patient-yrs. First postoperative year is marked by a 24% incidence of thrombosis. Stable incidence between the second to fourth years (~ 15%), and a subsequent decrease afterward. Mortality rates of Re-do Surgery have been reported to be from 6% to 69% (average 12%) Thrombolytic therapy as a First-line strategy is being used with successful outcomes. To Study the Efficacy & Safety of Low Dose (25 mg) Ultra-slow (24 hr) Infusion of Alteplase Without Bolus (max 72 hrs) over Slow (24hr) Infusion of 25 lac units Streptokinase (2.5 lac 1st hr → 1 lac /hr for 23 hrs) (max 48 hrs) in Mechanical PVT.

Objectives :

Primary :

To compare the success rate of USLD Alteplase thrombolysis over Streptokinase To compare the complication rates (minor + non-fatal major + fatal) in both the study groups

Secondary:

To study the clinical profile of patients presenting with Mechanical PVT. Single Centre Open Label Randomized Controlled Trial Sample Size : 100 (50 each) Follow up : Till Hospital Discharge Pt randomized as per Computer Generated Random Number Started on Inj Heparin Infusion till initiation of Thrombolysis. Repeat 2D Echo at 6 Hrs, 12 Hrs and 24 Hrs Interval & as required. Repeat Fluoroscopy / TEE if Echocardiographic evidence of improvement in gradient or moving leaflets / at 24 hrs interval.

Extended Thrombolysis with STK (max 48 hrs) / Alteplase (Max 72 hrs) Restarting of Heparin Infusion In between time lags for next continuation of Thrombolysis / Surgery/ attaining Therapeutic INR Post-thrombolysis Follow up till Discharge for Outcome

ELIGIBILITY:
patients with Written Informed Consent All adult patients of Mechanical PVT, Patient planned for Thrombolysis as first option as per common decision of Treating Cardiologist and CVTS Team.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
complication rates | 30 days
  To compare the success rate of USLD Alteplase thrombolysis over Streptokinase To compare the complication rates (minor + non-fatal major + fatal) in both the study groups

CONTACTS AND LOCATIONS:
Overall Officials: Sibasis Sahoo, DM, Principal Investigator — U. N. Mehta Institute of Cardiology and Research Center
Locations (1):
- Dr.Sibasis Sahoo, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No
Patients information don't want to disclose